CLINICAL TRIAL: NCT04351659
Title: Novel Adoptive Cellular Therapy With SARS-CoV-2 Specific T Cells in Patients With Severe COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singapore General Hospital (Other); National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-T 1.0
Record Dates: First submitted 2020-04-16; First posted 2020-04-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Coronavirus disease
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood from COVID-19 convalescent donors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood donors: Donors who had tested positive for SARS-CoV-2 in the past and have recovered from COVID-19 and are now suitable for blood donation.
  Interventions: Other: Blood donation from convalescent donor

INTERVENTIONS:
Other: Blood donation from convalescent donor — Donation of 1 unit of blood or leukapheresis

SUMMARY:
The overall objective of this project is to develop an emergent treatment protocol using adoptive T-cell therapy for the treatment of severe COVID-19. The central hypothesis is that SARS-CoV-2 specific T cells from convalescent donors who have recovered from COVID-19 can be manufactured expeditiously for the treatment of severe SARS-CoV-2 infections.

DETAILED DESCRIPTION:
A novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the cause of Coronavirus Disease 2019 (COVID-19). Currently, no vaccine or specific treatment has been proven to be effective. While waiting for vaccine to be developed, passive immunity can be acquired immediately by adoptive transfer of SARS-CoV-2 specific T cells from convalescent donors into newly infected patients.

The aim of this protocol is to demonstrate the feasibility of preparing SARS-CoV-2 specific T cells from convalescent donors for urgent clinical use. The specific hypothesis is that SARS-CoV-2 specific T cells can be isolated from the blood of convalescent donors rapidly and efficiently using SARS-CoV-2 specific peptides and an automated medical device for emergent treatment of severe COVID-19 disease.

A minimum of 8 convalescent donors will be recruited from Singapore to attain HLA sharing with at least 90% of the general population.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 65
* Had a history of COVID-19 with documented positive test for SARS-CoV-2 in the past
* Has recovered from COVID-19 and is now suitable for blood donation, fulfilling all standard blood donor criteria
* Negative test for SARS-CoV-2 currently

Exclusion Criteria:

* Do not meet the standard criteria for blood cell donation at National University Hospital or Singapore General Hospital.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential donors are those who have recovered from COVID-19 and are willing to donate blood for other COVID-19 patients.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Success rate in production of SARS-CoV-2 specific T cells from convalescent donor | Two weeks (The expected duration of donor participation is 2 weeks)
  Success of SARS-CoV-2 specific T cell manufacturing is defined as production of >200,000 T cells per donor. The success rate will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Wing Hang Leung, Principal Investigator — KK Hospital, SingHealth, Duke-NUS
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore